CLINICAL TRIAL: NCT04809493
Title: Evaluation of the Effect of Isonatremic (vs Conventional) Dialysis Treatment on the Control of Interdialytic Weight Gain in Chronic Kidney Disease Patients on Dialysis (Stage 5D)
Brief Title: Study Evaluating the Effect of Isonatremic Dialysis Treatment in Chronic Kidney Disease Patients on Dialysis
Acronym: DISON-IRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0659
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease patient on dialysis (stage 5D); Extracorporeal purification; Isonatremic dialysis; Sodium
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients will be receiving conventional dialysis: Patients will be receiving conventional dialysis treatment followed by isonatremic dialysis treatment during an observational period of 2 months for each treatment
  Interventions: Procedure: Conventional dialysis treatment; Procedure: Isonatremic dialysis treatment

INTERVENTIONS:
Procedure: Conventional dialysis treatment — Conventional dialysis treatment
Procedure: Isonatremic dialysis treatment — Isonatremic dialysis treatment

SUMMARY:
Aim of this study is to evaluate, in a population of chronic kidney disease patients on dialysis (Stage 5D), the effect of treatment with isonatremic dialysis (vs conventional dialysis), during an observational period of 2 months each, on:

* control of interdialytic weight gain
* perdialytic tolerance in terms of adverse events occurring during all of the sessions of the study
* body composition and thirst measured monthly during the 4 months of follow-up.
* tolerance to treatment.

ELIGIBILITY:
Inclusion criteria:

* Chronic Kidney Disease patient on dialysis (stage 5D)
* With plasma sodium concentration between 130 and 140 mmol/L
* Anuric
* Patient dialysed with dialysis machine allowing isonatremic dialysis treatment

Exclusion criteria:

* Patient with plasma sodium concentration below 130 or above 140 mmol/
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients issued from dialysis units (hospital, clinic, non profit dialysis centers)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of interdialytic weight gain during treatment | 1, 2, 3 and 4 months after inclusion
  change of interdialytic weight gain during treatment with isonatremic dialysis vs conventional dialysis during an observational period of 2 months each one.

SECONDARY OUTCOMES:
Perdialytic tolerance in terms of adverse events occurring | 1, 2, 3 and 4 months after inclusion
  Perdialytic tolerance in terms of adverse events occurring during all sessions of the study with isonatremic dialysis vs conventional dialysis for an observational period of 2 months each one.
Body composition | 1, 2, 3 and 4 months after inclusion
  Body composition monthly during treatment with isonatremic dialysis vs conventional dialysis during an observational period of 2 months each one.
Rate of Tolerance | 1, 2, 3 and 4 months after inclusion
  Rate of Tolerance during treatment with isonatremic dialysis vs conventional dialysis during an observational period of 2 months each one.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Study Director — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC